CLINICAL TRIAL: NCT03103711
Title: A Brief Psychological Intervention Using Virtual Reality for the Promotion of Emotional Well-being in Hospitalized Cancer Patients
Brief Title: Promotion of Emotional Well-being in Hospitalized Cancer Patients by Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Hospital Clínica Benidorm (Unknown); Universitat Jaume I (Other); Universitat Politècnica de València (Other)
Responsible Party: Principal Investigator, Rosa María Baños Rivera, Full Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONCOTIC-I
Record Dates: First submitted 2017-03-21; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Cancer
Keywords: Virtual reality; Well-being; Hospital
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The entire intervention is composed by four 30 minutes sessions along 1 week. Its focus is on the promotion of well-being by the use of two virtual environments ("Emotional Parks" and "Walk through Nature"). These environments allow participants to involve in different exercises (working with self statements, videos, images, slow breathing, focus on the present exercises) with the purpose of increase positive emotional states.
  Interventions: Behavioral: Virtual Reality Intervention
- Control (No Intervention): Participants receive the medical treatment deliver by the hospital. They fulfill several questionnaires at two moments (pre and post 1 week after). After this, they have the possibility to receive the psychological intervention.

INTERVENTIONS:
Behavioral: Virtual Reality Intervention — Participants receive two sessions oriented to joy and two focused on relax. In the first 2 sessions patients can choose the environment ("Emotional Parks" or "Walk through Nature") and in the following ones participants visit the alternate environments.
  Arms: Intervention

SUMMARY:
The aim of this study is to analyze the effect of a brief psychological intervention supported by Information and Communication Technologies, on the subjective well-being of hospitalized cancer patients. Participants are randomly assigned to one of 2 conditions: Intervention condition (4 Virtual reality sessions) and Control condition (waiting list control group).

ELIGIBILITY:
Inclusion Criteria:

* adults with any cancer diagnosis
* hospitalized for at least 1 week
* Karnofsky functional state ≥50
* life expectancy ≥2 months

Exclusion Criteria:

* serious psychopathology
* cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983; adapted version of Tejero, Guimerá, Farré & Peri, 1986) | change from baseline at 1 week
Fordyce Happiness Scale (Fordyce, 1988). | change from baseline at 1 week

SECONDARY OUTCOMES:
Visual Analog Scale: Mood. | 4 days along 1 week
  Subjective mood change after each intervention session.
Visual Analog Scale: Emotional State. Change from pre to post session. | 4 days along 1 week
  Assessment of general mood, joy, sadness, anxiety, relax and vigor (7-point Likert scale)
Visual Analog Scale: Physical Discomfort. Change from pre to post session. | 4 days along 1 week
  Presence of pain, fatigue and physical discomfort (11-point Likert scale)
Visual Analog Scale: Satisfaction with the Session Scale. | 4 days along 1 week
  Level of pleasantness and perceived usefulness of each session (11-point Likert scale)
Satisfaction with Intervention Scale (adapted version of Borkovec and Nau's, 1972) | 1 week
  Assesses satisfaction, recommendation, utility and discomfort (11-point Likert scale)

OTHER OUTCOMES:
The Brief Illness Perception Questionnaire (BIPQ) (Broadbent et al., 2006) | baseline
  This instrument has 9 items aimed to evaluate the cognitive and emotional representation of the illness (consequences, timeline, personal control, treatment control, identity, concern, emotional response, illness coherence and causes).
Personal meaning of the illness (ad-hoc). | baseline
  Patient has 6 alternatives of illness meaning (Loss, threat, challenge, blame-others, blame-self and opportunity). In addition to these alternatives, participant can add any other personal meaning.
Visual Analog Scale: Optimism | baseline
  11-point scale (not at all - completely)
Visual Analog Scale: Life satisfaction | baseline
  7-point scale (no satisfaction - completely satisfied)